CLINICAL TRIAL: NCT06377254
Title: Concurrent Multi-organ Responses to CHronic Physical Activity and INactivity Intervention, to Increase Research Discovery in Human Health and Wellbeing
Brief Title: Multi-organ Responses to CHronic Physical Activity and INactivity
Acronym: CHAIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Biotechnology and Biological Sciences Research Council (Other)
Responsible Party: Principal Investigator, Paul Greenhaff, Principal Investigator, University of Nottingham
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: BB/X015173/1
Record Dates: First submitted 2024-04-11; First posted 2024-04-22 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Sedentary Behavior; Metabolic Syndrome; Age-related Cognitive Decline; Age-Related Sarcopenia
Keywords: Physical activity; middle-age; Physical inactivity; overweight; lifestyle
MeSH Terms: conditions — Sedentary Behavior; Metabolic Syndrome; Motor Activity; Overweight

STUDY DESIGN:
Intervention Model Description: Non-randomised, parallel design lifestyle intervention
Who Masked: Outcomes Assessor
Masking Description: Those undertaking analysis of biological samples and MRI data will be masked as to the group the participant is allocated to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inactivity (Experimental): Participants in this group will reduce their physical activity (increase sitting time to 7hrs/day and decrease step count to <4500/day) for 3 months, then increase their activity for 3 months, through attending 3x 45 min supervised exercise sessions/week.
  Interventions: Behavioral: Decreased Physical Activity
- Activity (Experimental): Participants in this group will have moderate intensity physical activity levels increased for 6 months, through attending 3x 45 min supervised exercise sessions/week.
  Interventions: Behavioral: Increased Physical activity

INTERVENTIONS:
Behavioral: Decreased Physical Activity — Physical activity levels will be decreased
  Arms: Inactivity
Behavioral: Increased Physical activity — Physical activity levels will be increased
  Arms: Activity

SUMMARY:
Life expectancy has been increasing for the last 150 years, but the maintenance of health has not kept pace with increased lifespan, and on average, UK adults spend the last decade of life in poor-health, with major consequences for society and the individual.

Persistent physical inactivity is thought to be a key contributing factor to the risk of poor health and functional decline occurring in middle-aged and older adults. It is therefore concerning that most middle-aged adults spend >8hrs/day being sedentary, with average step count of 3000-4000 steps/day.

To be able to holistically assess the effectiveness of future strategies to address age-related decline in health, and devise public health messages to help individuals reach older age in better health, it is essential that the complex physiological effects that activity and inactivity have across biological systems are characterised.

The goal of this intervention study is to compare the impact of physical activity and inactivity on body functioning. Twenty moderately active participants will decrease their physical activity for three months to match the average amount carried out by middle-aged people in the UK. They will then undertake 3-months of reconditioning training to restore their fitness. In addition, twenty sedentary participants will increase their physical activity to UK recommended levels for six months.

Before and at points during the intervention period, participants will be asked to make some measurements at home and attend the University of Nottingham to have multiple assessments made. These include;

* fitness, muscle strength and function tests,
* completion of questionnaires and computer-based brain puzzles
* having muscle and fat tissue biopsies and blood samples taken.
* The study also involves having MRI scans.

This 5-year study will commence in January 2024, with participant recruitment starting in March 2024 and finishing in May 2027.

DETAILED DESCRIPTION:
This is a parallel design study comparing the impact of physical activity and inactivity on the way the body functions, to understand the mechanisms (including the inter-relationship between tissues and organs) by which lifestyle behaviours may effect health and wellbeing in later life. In particular, the mechanisms by which inactivity results in long term poor health is not well understood, and has rarely been studied in an integrated way in people. However, initial research indicates that the physiology of being inactive is not simply the reverse of being active. To enable effective treatments and public health advice to be devised so that more adults reach old age in better health, and maintain a good quality of life for a greater proportion of their older age, it is important that the impact of physical inactivity on the way the body functions is better understood. Therefore, twenty participants who are moderately, but not highly active will be asked to decrease their physical activity for three months to match the average exercise levels of middle-aged people in the United Kingdom (UK). This will require them to increase their daily sitting time to 7 hours a day and reduce their step count to <4500 steps per day. At the end of the 3-months they will undertake 3-months of supervised reconditioning training by attending the Medical School at Queen's Medical Centre, Nottingham, three times a week.

In addition, twenty participants who currently have low physical activity levels will be asked to increase their physical activity to UK recommended levels by attending the Medical School at Queen's Medical Centre, Nottingham, three times a week for six months to undertake a supervised exercise program.

Before and during the 6-month period (at weeks 6, 12, 18 and 24) participants will be asked to make some measurements at home (physical activity levels, dietary intake) and attend the University of Nottingham over 4 days to have multiple assessments made. These include: height; weight; body composition (body fat and lean tissue); blood pressure; fitness, muscle strength and function; sleep quality, quality of life and wellbeing (questionnaires). The rate of muscle protein breakdown and muscle protein synthesis, blood sugar regulation, and biochemistry of the blood, fat tissue and muscles will be assessed, and to enable this muscle and fat tissue biopsies will be collected and blood samples taken. The study also involves having MRI scans to study the structure and function of the brain and heart, and to determine liver and muscle fat content.

ELIGIBILITY:
Inclusion Criteria:

* Group 1 ('non-sedentary') self-reporting <6 sedentary hrs/day, not actively involved in exercise training or a regular physical activity regimen (>8,000 steps/day).
* Group 2 ('sedentary') self-reporting ≥8 waking hrs/day in sedentary activities and/or ≤5,000 steps/day.
* Aged 50-65y.
* Overweight (BMI 25-35 kg/m2).
* Waist circumference ≥94cm (males) and ≥80cm (females).
* Willing to alter physical activity levels as instructed for 6 months
* Without neurological or psychiatric diseases, motor or cognitive restrictions
* Ability to give informed consent

Exclusion Criteria:

* Regular medication use that could interfere with measures
* A history, or evidence, of chronic cardiovascular, metabolic, musculoskeletal, renal or respiratory diseases.
* Experiencing 'long-COVID', inflammatory bowel disease or malignancy.
* Uncontrolled hypertension. Stage 1 hypertension (BP ≤160/100mmHg) with no other signs of cardiovascular disease, and blood pressure (BP) managed by routine medication will not be an exclusion.
* People employed in jobs that would preclude reducing step count and night-shift workers.
* Females who are pre/peri-menopausal, (due to effect of oestrogen fluctuations on primary outcomes and the longitudinal study design), but individuals stable on hormone replacement therapy are eligible.
* Contraindications for MRI.
* Allergy or sensitivity to local anaesthesia, or dressing adhesive

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2027-12-17 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in Cardiorespiratory fitness (VO2 max) | 12 weeks
  change in maximal oxygen uptake (continuous incremental bicycle ergometer exercise test with on-line gas analysis) measured every 6 weeks

SECONDARY OUTCOMES:
Change in Isometric leg strength | 24 weeks
  Change in Isometric leg strength measured every 6 weeks using CYBEX dynamometer
Change in time to leg fatigue | 24 weeks
  Change in time taken to induce muscle fatigue measured every 6 weeks using isokinetic knee extensions on a CYBEX dynamometer
Change in incremental area under the curve (iAUC) for blood glucose concentration | 24 weeks
  Change in 180 minute blood glucose concentration incremental area under the curve measured every 6 weeks during an oral glucose tolerance test.
Change in iAUC for serum insulin concentration | 24 weeks
  Change in 180-minute serum insulin concentration incremental area under the curve measured every 6 weeks during an oral glucose tolerance test
Change in fasting glucose oxidation rate | 24 weeks
  Change in glucose oxidation rate (when fasted), measured every 6 weeks using ventilated hood indirect calorimetry
Change in 'fed' glucose oxidation rate | 24 weeks
  Change in glucose oxidation rate (in the insulin-stimulated 'fed' state), measured every 6 weeks using ventilated hood indirect calorimetry during an oral glucose tolerance test
Change in Short Form Health Survey (SF36) Questionnaire aggregated normalised 'physical' score | 24 weeks
  Change in 'SF36' Questionnaire aggregated 'physical' score (normalised to UK population) calculated according to standard procedures (min 0, max 100), with higher score indicating better physical wellbeing measured every 6 weeks
Change in Short Form Health Survey (SF36) Questionnaire aggregated and normalised 'mental' score | 24 weeks
  Change in 'SF36' Questionnaire aggregated 'mental' score (normalised to UK population) calculated according to standard procedures (min 0, max 100), with higher score indicating better mental wellbeing, measured every 6 weeks
Change in World Health Organisation Quality of Life (WHOQoL) score | 24 weeks
  Change in World Health Organisation Quality of Life Score (measured using the WHOQoL-Bref questionnaire every 6 weeks), (min score 0, max 100), with higher score indicating a better state of health.
Change in Pittsburgh Sleep Quality Index (PSQI) | 24 weeks
  Change in PSQI score (min score 0, max 21), measured every 6 weeks, with higher score indicating poorer sleep quality
Change in Stroop test; % Accuracy | 24 weeks
  Change in the percentage of accurate responses, measured every 6 weeks, with higher score indicating better cognitive performance. Minimum value 0%, maximum value 100%
Change in Stroop test; reaction time | 24 weeks
  Change in the reaction time for responses, measured every 6 weeks, with higher score indicating slower cognitive performance. No minimum or maximum value defined.
Change in four-choice reaction time test; % Accuracy | 24 weeks
  Change in the percentage of accurate responses, measured every 6 weeks, with higher score indicating better cognitive performance. Minimum value 0%, maximum value 100%
Change in four-choice reaction time test; reaction time | 24 weeks
  Change in the reaction time for responses, measured every 6 weeks, with higher score indicating slower cognitive performance. No minimum or maximum value defined.
Change in card sort test; % Accuracy | 24 weeks
  Change in the percentage of accurate responses, measured every 6 weeks, with higher score indicating better cognitive performance. Minimum value 0%, maximum value 100%
Change in card sort test; reaction time | 24 weeks
  Change in the reaction time for responses, measured every 6 weeks, with higher score indicating slower cognitive performance. No minimum or maximum value defined.
Change in Logical reasoning test; % accuracy | 24 weeks
  Change in the accuracy of responses, measured every 6 weeks, with higher score indicating better cognitive performance. Minimum value 0%, maximum value 100%
Change in Logical reasoning test; reaction time | 24 weeks
  Change in the reaction time for responses, measured every 6 weeks, with higher score indicating slower cognitive performance. No minimum or maximum value defined.
Change in serial subtractions test; number of responses in 2 minutes | 24 weeks
  Change in the number of responses, measured every 6 weeks, with higher score indicating better cognitive performance. minimum number is 0, maximum number is variable dependent on starting value (800-999; randomly selected by computer program) and speed of response.
Change in Corsi blocks test; score | 24 weeks
  Change in the test score, measured every 6 weeks, with higher score indicating better cognitive performance.Minimum score is 0 and maximum is 15.
Change in Muscle protein synthesis rate | 24 weeks
  Muscle synthesis protein rate calculated from deuterium incorporation into muscle tissue
Change in Muscle protein breakdown rate | 24 weeks
  Muscle protein breakdown rate calculated every 6 weeks using 3-methylhistidine tracer
Change in whole body fat volumes | 24 weeks
  Change in the amount of fat within the body, measured every 6 weeks using magnetic resonance imaging (MRI)
Change in liver fat volumes | 24 weeks
  Change in the amount of fat within the liver, measured every 6 weeks using magnetic resonance imaging (MRI)
Change in thigh muscle fat volumes | 24 weeks
  Change in the amount of fat within the vastus lateralis thigh muscle, measured every 6 weeks using magnetic resonance imaging (MRI)
Change in whole body muscle volumes | 24 weeks
  Change in the amount of muscle within the body, measured every 6 weeks using magnetic resonance imaging (MRI)
Change in muscle phosphocreatine synthesis rate | 24 weeks
  Change in the rate of phosphocreatine synthesis, measured every 6 weeks using magnetic resonance spectroscopy
Change in cerebral volume | 24 weeks
  Change in the volume of brain tissue, measured every 6 weeks using magnetic resonance imaging (MRI)
Change in cortical thickness | 24 weeks
  Change in the thickness of the brain cortex, measured every 6 weeks using magnetic resonance imaging (MRI)
Change in plasma metabolome | 24 weeks
  change in untargeted plasma metabolome profile measured every 6 weeks

OTHER OUTCOMES:
Fasting blood lipid concentration | pre-intervention
  concentration of lipid within the blood
Fasting blood lipid concentration | 6 weeks
  concentration of lipid within the blood
Fasting blood lipid concentration | 12 weeks
  concentration of lipid within the blood
Fasting blood lipid concentration | 18 weeks
  concentration of lipid within the blood
Fasting blood lipid concentration | 24 weeks
  concentration of lipid within the blood
liver function test: alanine transaminase (ALT) | pre-intervention
  concentration of ALT measured on blood sample
liver function test: alanine transaminase (ALT) | 6 weeks
  concentration of ALT measured on blood sample
liver function test: alanine transaminase (ALT) | 12 weeks
  concentration of ALT measured on blood sample
liver function test: alanine transaminase (ALT) | 18 weeks
  concentration of ALT measured on blood sample
liver function test: alanine transaminase (ALT) | 24 weeks
  concentration of ALT measured on blood sample
liver function test: aspartate aminotransferase (AST) | pre-intervention
  concentration of AST measured on blood sample
liver function test: aspartate aminotransferase (AST) | 6 weeks
  concentration of AST measured on blood sample
liver function test: aspartate aminotransferase (AST) | 12 weeks
  concentration of AST measured on blood sample
liver function test: aspartate aminotransferase (AST) | 18 weeks
  concentration of AST measured on blood sample
liver function test: aspartate aminotransferase (AST) | 24 weeks
  concentration of AST measured on blood sample
liver function test: Bilirubin | pre-intervention
  concentration of bilirubin measured on blood sample
liver function test: Bilirubin | 6 weeks
  concentration of bilirubin measured on blood sample
liver function test: Bilirubin | 12 weeks
  concentration of bilirubin measured on blood sample
liver function test: Bilirubin | 18 weeks
  concentration of bilirubin measured on blood sample
liver function test: Bilirubin | 24 weeks
  concentration of bilirubin measured on blood sample
liver function test: Albumin | pre-intervention
  concentration of albumin measured on blood sample
liver function test: Albumin | 6 weeks
  concentration of albumin measured on blood sample
liver function test: Albumin | 12 weeks
  concentration of albumin measured on blood sample
liver function test: Albumin | 18 weeks
  concentration of albumin measured on blood sample
liver function test: Albumin | 24 weeks
  concentration of albumin measured on blood sample
liver function test: Gamma glutamyl transferase (GGT) | pre-intervention
  concentration of GGT measured on blood sample
liver function test: Gamma glutamyl transferase (GGT) | 6 weeks
  concentration of GGT measured on blood sample
liver function test: Gamma glutamyl transferase (GGT) | 12 weeks
  concentration of GGT measured on blood sample
liver function test: Gamma glutamyl transferase (GGT) | 18 weeks
  concentration of GGT measured on blood sample
liver function test: Gamma glutamyl transferase (GGT) | 24 weeks
  concentration of GGT measured on blood sample
Blood Haemoglobin concentration | pre intervention
  haemoglobin concentration measured on a blood sample
Blood Haemoglobin concentration | 6 weeks
  haemoglobin concentration measured on a blood sample
Blood Haemoglobin concentration | 12 weeks
  haemoglobin concentration measured on a blood sample
Blood Haemoglobin concentration | 18 weeks
  haemoglobin concentration measured on a blood sample
Blood Haemoglobin concentration | 24 weeks
  haemoglobin concentration measured on a blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Paul L Greenhaff, PhD, Principal Investigator — University of Nottingham
Locations (1):
- David Greenfield Human Physiology Unit, Nottingham, Notts, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised dataset will be made available to other researchers on request after study aims have been analysed and published. No patient identifiable data will be shared
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will become available approximately 2 years after study completion and will be available for 20 years
Access Criteria: Although parts of the data set generated from this project will be available on open access platforms to support publications, access to the full data repository and tissue archive will be through requests made to the Management Board. Access will be subject to ethical constraints, the preservation of intellectual property (IP), and written acknowledgement that it is a research collaboration, with data ownership residing with the original research teams. Data will be shared subject to a data transfer agreement and confirmation that deletion of the shared data set will occur once analysis has been completed.